CLINICAL TRIAL: NCT00325767
Title: Mucociliary Clearance in Healthy Subjects: Comparison of Levalbuterol and Racemic Albuterol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RPN 04-03-19-11
Record Dates: First submitted 2006-05-12; First posted 2006-05-15 (Estimated); Last update posted 2006-05-15 (Estimated); Status verified 2006-04

CONDITIONS: Mucociliary Clearance
Keywords: mucociliary clearance; beta-adrenergic drugs; inhalation; aerosol
MeSH Terms: conditions — Respiratory Aspiration

INTERVENTIONS:
Drug: nebulized albuterol (2.5 mg/3ml/dose)
Drug: nebulized levalbuterol (1.25 mg/3ml/dose)
Drug: nebulized placebo (3ml/dose)

SUMMARY:
The purpose of this study is to determine whether lung mucociliary clearance (MCC) can be significantly enhanced in healthy subjects by one week of inhalation of nebulized levalbuterol aerosol, as compared to racemic albuterol or placebo. Subjects will inhale one week of levalbuterol, one week of racemic albuterol, and one week of placebo, in a randomized order.

DETAILED DESCRIPTION:
In healthy lungs, inhaled insoluble material such as bacteria, viruses, antigens, and toxins deposit in the tracheobronchial airway mucus and are removed from the lung in a matter of hours by mucociliary clearance (MCC). When MCC is overwhelmed or impaired, some mucus can be removed by mechanical or cough clearance (CC). Impairment of MCC typically leads to the accumulation of mucus in the airways, and this in turn is associated with acute infections, chronic bacterial colonization, and chronic inflammation.

Racemic albuterol has been shown to stimulate MCC in various patient populations. Inhaled and subcutaneous terbutaline has also been shown to stimulate MCC in healthy subjects. We hypothesize that levalbuterol will be more potent than racemic albuterol in enhancing MCC and CC in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* non-smoking males and non-pregnant females greater than or equal to 18 years of age
* forced expiratory volume in one second (FEV1) and forced vital capacity (FVC) greater than or equal to 80% of predicted values
* normal systolic and diastolic blood pressures

Exclusion Criteria:

* history of heart disease, irregular heartbeat, hypertension
* history of diabetes, hyperthyroid
* history of pneumonia, tuberculosis
* history of seizure disorder, depression, hospitalization in the last month for non-elective purposes, cold or flu in the previous three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2004-05; Study Completion 2005-09

PRIMARY OUTCOMES:
Lung mucociliary clearance
Lung cough clearance

SECONDARY OUTCOMES:
Forced expiratory volume in 1 second
Forced vital capacity

CONTACTS AND LOCATIONS:
Overall Officials: Beth L Laube, Ph.D., Study Director — Johns Hopkins University; Jeffrey C Cleary, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Eudowood Division of Pediatric Respiratory Sciences, Baltimore, Maryland, United States